CLINICAL TRIAL: NCT02770638
Title: A Comparison of Tissue Interface Pressures and Comfort Ratings of the Scoop Stretcher and Traditional Long Back Board in Rugby and University Athletes
Brief Title: Tissue Interface Pressures in Athlete Medical Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Kimberley Edwards, Professor Sport Exercise & Nutrition Education, University of Nottingham
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: G10042014 SoM ROD
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Emergency; Pain; Medical Device Discomfort
Keywords: Healthy; Sport; Athlete; Male; University; Adults; Rugby Football Union; Professional; Competitive sport; Scoop Stretcher; Ferno Scoop Stretcher; Long back spinal board; Emergency Medical Services; Long backboard; Patient Extrication; Triple Immobilisation; Pre hospital Medicine; Rigid Cervical Collar; Pressure Testing; Tissue Pressure Testing; Visual Analogue Scale; Pressure Sores; Pressure area damage; Tissue Viability; Tissue Interface Pressure; Comfort; Pain
MeSH Terms: conditions — Emergencies; Pain; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scoop Stretcher (Experimental): Participant wearing light sports clothing will start with forty five minutes laid supine on the scoop stretcher with 'triple immobilisation ' (rigid cervical collar, two headblocks and fastening straps). Followed by a forty five minute washout period (participant can mobilise freely). Participants will complete the observation with forty five minutes laid supine on the long back spinal board with 'triple immobilisation ' (rigid cervical collar, two headblocks and fastening straps).
  Interventions: Device: Scoop Stretcher
- Long Back Spinal Board (Active Comparator): Participant wearing light sports clothing will start with forty five minutes laid supine on the long back spinal board with 'triple immobilisation ' (rigid cervical collar, two headblocks and fastening straps). Followed by a forty five minute washout period (participant can mobilise freely). Participants will complete the observation with forty five minutes laid supine on the scoop stretcher with 'triple immobilisation ' (rigid cervical collar, two headblocks and fastening straps).
  Interventions: Device: Long Back Spinal board

INTERVENTIONS:
Device: Scoop Stretcher — Participants recruited by community advertisement. Participant will complete forty five minutes on scoop stretcher first, followed by forty five minute washout period, finished with forty five minutes on the long back spinal board. Tissue pressures will be automatically recorded throughout the forty five minute period laid on either spinal board. In addition, participants will be asked to report their comfort levels at five minute intervals.
  Other Names: Trade Name: Ferno Scoop Stretcher
  Arms: Scoop Stretcher
Device: Long Back Spinal board — Participants recruited by community advertisement. Participant will complete forty five minutes on the long back spinal board first, followed by forty five minute washout period, finished with forty five minutes on the scoop stretcher. Tissue pressures will be automatically recorded throughout the forty five minute period laid on either spinal board. In addition, participants will be asked to report their comfort levels at five minute intervals.
  Arms: Long Back Spinal Board

SUMMARY:
This study aims to establish clinical evidence for the use of scoop stretchers in the sports setting for spinal immobilisation and transport compared to the traditionally used long back boards through measuring tissue interface pressures over forty five minutes. All participants will be placed on both the scoop stretcher and the long back board for forty five minutes each, with at least 45 minutes between the two tests. A special mat that measures the pressure of the body against the board will be used to determine the pressure forces at certain points of the body touching the board (in mmHg). The participants will also be asked every five minutes during the experiment to rate the comfort of the device. Pressure measures from each participant on each board will be collated and assessed along with each participant's reported pain scores and comfort rating. The measurements from the tissue pressures will be analysed in real-time from the software connected to the pressure-mat and therefore show if pressures increase over time. A comparison between boards will be made.

DETAILED DESCRIPTION:
Background

In recent years the scoop stretcher, for a number of reasons, has been advocated by the Faculty for Pre-hospital Care (Royal College of Surgeons Edinburgh, United Kingdom) as the 'Gold Standard' method of extrication and transport in pre-hospital trauma and this has been extrapolated to extricating athletes from the field of play in sport who have sustained a potential spine injury. In addition they have advised that the conventional long back boards should no longer to be used as a stretcher, only a pure extrication device. This has an implication to the emergency care currently provided in sport and will affect every sports club financially and every medical team who require training in the use of the new device.

Previous research studies have looked at how much pressure lying on different spinal boards (e.g. the long back board or vacuum mattress) causes the athlete. This is because of a concern that lying on a board for too long may cause pressure sores or other medical complications. However, no research has been done to measure these tissue pressures using the scoop stretcher which is now indicated for general use in pre-hospital care in sport. Also there is no evidence to compare how comfortable athletes find the different spinal boards.

Aims

This observational study aims to measure the tissue interface pressures and perceived levels of comfort of rugby players and University participants (staff and students) immobilised on a scoop stretcher and on a long back board for forty five minutes. It will also enable the changes in pressures and comfort ratings over time to be assessed to evaluate the appropriate time cut off for such immobilisation.

Experimental Protocol and Methods

A prospective cross-over study. Players from Nottingham Rugby Football Club and the University of Nottingham (staff and students) will be invited to participate for the study (summer 2016). Participants will be randomly (block randomisation) assigned to start on either the scoop or long board. Participants will be log rolled onto each board and fully immobilised for forty five minutes. The wash out period will be a minimum of forty five minutes. All measurements will be collected on the same pressure mat.

Measureable end points/statistical power of the study

The pressure mat (provided by BES Rehab) will be laid on top of the spinal board and will automatically measure the tissue interface pressure readings (occiput, scapulae, sacrum, heels) every five minutes. Participant reported pain will be measured by a Visual Analogue Scale (VAS) and will be used to collect the comfort ratings data (occiput, scapulae, sacrum, heels, overall) every five minutes. Age, height, weight, sport team and position played and length of sporting participation will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, uninjured - no current sports injury, male, 75kg (165 lb) in weight or over.

Exclusion Criteria:

* Female, weight less than 75kg (165 lb)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Occiput tissue pressure in millimetres mercury (mmHg) | 1 day

SECONDARY OUTCOMES:
Scapulae tissue pressure in millimetres mercury (mmHg) | 1 day
Sacrum tissue pressure in millimetres mercury (mmHg) | 1 day
Heels tissue pressure in millimetres mercury (mmHg) | 1 day
Subjective participant reported pain levels using visual analogue scale (VAS) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley L Edwards, MMedSci PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanson JR, Carlin B. Sports prehospital-immediate care and spinal injury: not a car crash in sight. Br J Sports Med. 2012 Dec;46(16):1097-101. doi: 10.1136/bjsports-2012-091800. Epub 2012 Oct 18. PMID 23080314
- [Background] Krell JM, McCoy MS, Sparto PJ, Fisher GL, Stoy WA, Hostler DP. Comparison of the Ferno Scoop Stretcher with the long backboard for spinal immobilization. Prehosp Emerg Care. 2006 Jan-Mar;10(1):46-51. doi: 10.1080/10903120500366375. PMID 16418091
- [Background] Moss R, Porter K, Greaves I; consensus group. Minimal patient handling: a faculty of prehospital care consensus statement. Emerg Med J. 2013 Dec;30(12):1065-6. doi: 10.1136/emermed-2013-203205. PMID 24232010